CLINICAL TRIAL: NCT02256761
Title: Safety, Pharmacokinetics, and Pharmacodynamics of BIRT 2584 XX Administered as Multiple Doses of 100 mg to 750 mg qd for 14 or 28 Days (Randomised, Double-blind Placebo Controlled Design), and Safety and Pharmacokinetics of 500 mg of BIRT 2584 XX Administered With and Without Food as Single Dose (Open, Intra-individual Comparison) to Healthy Male Volunteers
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of BIRT 2584 XX Administered as Multiple Doses and Safety and Pharmacokinetics of BIRT 2584 XX Administered With and Without Food as Single Dose to Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1206.2
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (3):
- BIRT 2584 XX - single dose (Experimental): Part 1 - bioavailability/food effect
  two single doses, 30 minutes prior to the second drug administration after a one week wash-out period, a standardised high fat, high caloric meal was served
  Interventions: Drug: BIRT 2584 XX - single dose; Other: high caloric meal
- Placebo (Placebo Comparator): Part 2
  Interventions: Drug: Placebo
- BIRT 2584 XX - multiple escalating dose (Experimental): Part 2 - multiple escalating dose, 14 days and 28 days
  Interventions: Drug: BIRT 2584 XX - multiple escalating dose

INTERVENTIONS:
Drug: BIRT 2584 XX - multiple escalating dose
  Arms: BIRT 2584 XX - multiple escalating dose
Drug: Placebo
  Arms: Placebo
Drug: BIRT 2584 XX - single dose
  Arms: BIRT 2584 XX - single dose
Other: high caloric meal — 30 minutes prior to the second drug administration after a one week wash-out period, a standardised high fat, high caloric meal was served
  Arms: BIRT 2584 XX - single dose

SUMMARY:
The study comprised two parts. The objective of the first study period was to assess the safety and pharmacokinetics of 500 mg of BIRT 2584 XX tablets administered with and without food in male healthy volunteers and to determine the relative bioavailability of the BIRT 2584 XX tablet formulation compared by historical comparison to BIRT 2584 XX powder in PEG 400 (U05-2074) (part 1). The second and major phase of the trial was aimed at evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple rising doses of BIRT 2584 XX (100 mg, 250 mg, and 500 mg bid on the first 2 days and qd on the following 12 days, or 750 mg qd for 28 days) in healthy male subjects (part 2)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of the screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age ≥ 18 and ≤ 63 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding during the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hematological, oncological, or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) considered relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (greater than 24 hours) (less than 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial (less than 10 days prior to study drug administration or expected during the trial)
* Participation in another trial with an investigational drug (less than 2 months prior to administration or expected during trial)
* Smoker (more than 10 cigarettes/day or more than 3 cigars/day or more than 3 pipes/day)
* Alcohol abuse (more than 60 g of ethanol per day)
* Drug abuse
* Blood donation or loss greater than 400 mL (less than 1 month prior to administration or expected during the trial)
* Clinically relevant laboratory abnormalities

Ages: 18 Years to 63 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2005-01; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal findings in physical examination | up to 45 days
Number of subjects with abnormal changes in laboratory parameters | up to 45 days
Number of subjects with clinically significant changes in vital signs | up to 45 days
  Pulse rate, systolic, and diastolic blood pressure
Number of subjects with adverse events | up to 59 days
Number of subjects with clinically significant changes in 12-lead ECG | up to 45 days

SECONDARY OUTCOMES:
AUC0-inf (area under the concentration-time curve of BIRT 2584 XX in plasma over the time interval from 0 to infinity) | up to 72 hours
  bioavailability/food effect part
Cmax (maximum concentration of BIRT 2584 XX in plasma) | up to 72 hours
  bioavailability/food effect part
tmax (time from dosing to maximum concentration of BIRT 2584 XX and BI 610100, its major metabolite in humans) | up to 72 hours
  bioavailability/food effect part
Cmax (maximum concentration of BIRT 2584 XX and BI 610100 in plasma) | up to 42 days
  multiple rising dose part
tmax (time from dosing to maximum concentration of BIRT 2584 XX and BI 610100) | up to 42 days
  multiple rising dose part
AUC0-12 (area under the concentration-time curve of BIRT 2584 XX and BI 610100 in plasma over the time interval from 0 to 12 hours after the first dose | up to 14 hours after first drug administration
  multiple rising dose part
AUCtau,l (area under the concentration-time curve of BIRT 2584 XX and BI 610100 in plasma over a uniform dose interval tau after administration of the last dose) | up to 42 days
  multiple rising dose part
Cmin,ss (minimum concentration of BIRT 2584 XX and BI 610100 in plasma at steady state over a uniform dosing interval tau) | up to 42 days
  multiple rising dose part
AUCtau,ss (area under the concentration-time curve of BIRT 2584 XX and BI 610100 in plasma at steady state over a uniform dosing interval tau) | up to 42 days
  multiple rising dose part
λz,ss (terminal rate constant of BIRT 2584 XX and BI 610100 in plasma at steady state) | up to 42 days
  multiple rising dose part
t1/2,ss (terminal half-life of BIRT 2584 XX and BI 610100 in plasma at steady state) | up to 42 days
  multiple rising dose part
MRTpo,ss (mean residence time of BIRT 2584 XX and BI 610100 in the body at steady state after po administration) | up to 42 days
  multiple rising dose part
CL/F,ss (apparent clearance of BIRT 2584 XX from plasma at steady state after extravascular multiple dose administration) | up to 42 days
  multiple rising dose part
Vz/F,ss (apparent volume of distribution of BIRT XX 2584 during the terminal phase λz at steady state following extravascular administration) | up to 42 days
  multiple rising dose part
Aet1-t2,ss (amount of BIRT 2584 XX and BI 610100 that is eliminated in urine at steady state from the time point t1 to time point t2) | up to 30 days
  multiple rising dose part
fet1-t2,ss (fraction of BIRT 2584 XX and BI 610100 eliminated in urine at steady state from time point t1 to the time point t2) | up to 30 days
  multiple rising dose part
Accumulation ratio of the analyte in plasma at steady state at the end of dosing expressed as a ratio of Cmax after the last dose to Cmax after the first dose (RA,Cmax) | up to 42 days
  multiple rising dose part
Accumulation ratio of the analyte in plasma at steady state at the end of dosing expressed as a ratio of AUCtau after the last dose to AUCtau after the first dose (RA,AUC) | up to 42 days
  multiple rising dose part
Assessment of receptor occupancy | up to 42 days
  determined by a competitive binding assay using anti-Lymphocyte function associated antigen-1 (LFA-1) antibody fragment as competitor
Assessment of ex vivo suppression of superantigen (SEB)-induced Interleukin (IL)-2 production | up to 42 days
Total number of white blood cells and leukocyte differential cell count | up to 42 days